CLINICAL TRIAL: NCT06723847
Title: Navigating the Learning Curve of Robotic Pancreatoduodenectomy: Feasibility, Proficiency, and Mastery in a First-generation Surgeon
Acronym: LC-RPD
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Niccolò Napoli, MD, PhD, FEBS, University of Pisa
Other Study IDs: LC-RPD-Boggi
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Robotic Pancreaticoduodenectomy
Keywords: learning curve; robotic pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — pancreatic head specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient underwent robotic pancreaticoduodenectomy: All patients undergoing robotic pancreaticoduodenectomy regardless of the pathology for which they underwent it
  Interventions: Procedure: Robotic pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Robotic pancreaticoduodenectomy — All procedures are performed used a standard technique of our center for robotic pancreaticoduodenectomy
  Other Names: robotic Whipple; robot-assisted pancreaticoduodenectomy; robot-assisted Whipple

SUMMARY:
This study delineates the learning curve of robotic pancreatoduodenectomy (RPD) for first-generation surgeons, using the Comprehensive Complication Index (CCI) to assess patient outcomes and the PD-ROBOSCORE to stratify patients for their risk to develop post-operative complications.

DETAILED DESCRIPTION:
This study aims to define the learning curve of a first-generation surgeon who implemented robotic pancreatoduodenectomy. When compared to previous studies on the same issue, the current study has several distinctive features. Firstly, the learning curve was defined using the cumulative sum method, with the comprehensive complication index as the main outcome metric. The comprehensive complication index provides a holistic view of the burden of postoperative complications in each individual patient, correlating with key outcome measures such as length of hospital stay, use of hospital resources, and ultimately mortality. Secondly, outcomes were adjusted by procedure complexity based on the newly described PD-ROBOSCORE (Surgery. 2023;173:1438-1446). This is the first study assessing the learning curve of robotic pancreatoduodenectomy while incorporating difficulty levels.

ELIGIBILITY:
Inclusion Criteria:

All patients underwent robotic pancreaticoduodenectomy.

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient underwent robotic pancreaticoduodenectomy at our institution regardless for the pathology
Sampling Method: Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Post-operative complications | 90 days
  90-day post-operative complications assessed by the Comprehensive Complication Index (CCI)

IPD SHARING:
Plan to Share IPD: No
They will be shared upon request